CLINICAL TRIAL: NCT02689323
Title: TMS Modulation of Insula-related Brain Networks
Acronym: TMS_INS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00069059
Record Dates: First submitted 2016-02-12; First posted 2016-02-23 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-04

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Experimental): Participants will undergo 5 sessions of active rTMS
  Interventions: Device: repeated transcranial magnetic stimulation

INTERVENTIONS:
Device: repeated transcranial magnetic stimulation

SUMMARY:
The purpose of this study is to investigate the modulatory effects of repetitive transcranial magnetic stimulation (rTMS) on functional connectivity with the insula. Functional connectivity (FC) measures the interaction between brain regions, and recent neuroimaging studies have used FC to investigate how addiction affects FC among pertinent brain regions. rTMS, which can excite cortical neurons, has shown promise as a method to manipulate brain connectivity and could be used therapeutically to treat addiction. However, investigators first need more information on brain FC and how it relates to behavior, in order to guide rTMS target selection.

ELIGIBILITY:
Inclusion Criteria:

1. generally healthy
2. between the ages of 18-55
3. right-handed

Exclusion Criteria:

1. significant health problems (e.g., current and uncontrolled liver, lung, or heart problems) or presence of medical illness likely to alter brain morphology (including history of seizure, history of epilepsy in self or first degree relatives, stroke, brain surgery, head injury, and known structural brain lesion)
2. current diagnosis of Axis I psychiatric disorders (e.g., depression, anxiety disorder, schizophrenia)
3. meet DSM-5 criteria for current substance use disorder other than nicotine
4. use of psychoactive medications that would result in a positive urine drug screen
5. Current use of medications known to lower the seizure threshold
6. positive breath alcohol concentration
7. presence of conditions that would make MRI unsafe (e.g., metal implants, pacemakers)
8. among women, a positive urine pregnancy test
9. vision that cannot be corrected to 20/40

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

PRIMARY OUTCOMES:
Change in functional connectivity strength measured with functional magnetic resonance imaging | baseline and 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No